CLINICAL TRIAL: NCT01336556
Title: Optimal Titration of Continuous Positive Airway Pressure Could Predict Success of Oral Appliance to Treat Obstructive Sleep Apnea Syndrome
Brief Title: Titration of Continuous Positive Airway Pressure Could Predict Success of Oral Appliance to Treat Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, professor, Associacao Fundo de Incentivo a Psicofarmcologia
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0352/09T
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral appliance; Continuous positive airway pressure; Obstructive Sleep Apnea Syndrome; Snore
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Oral appliance — Anterior mandibular repositioner: used for two months

SUMMARY:
Background: The oral appliances have been increasingly used in the treatment of primary snoring and in patients with mild obstructive sleep apnea syndrome besides being treatment options in adults with moderate to severe sleep apnea who did not accept or adapt to continuous positive airway pressure (CPAP). It is not well established yet in the literature, which patients with mild to moderate OSA will present a good response to treatment with oral appliances.

Objective: To determine a value of CPAP pressure that correlates with a favorable response to the use of oral appliance in patients with mild to moderate sleep apnea.

Patients and Methods: Two groups of 30 male patients (25-65 years, body mass index < 35 kg/m2) will be selected: the first group with an apnea-hypopnea index (AHI) between 5 and 15 events per hour of sleep and the second one with an AHI between 15 and 30 events per hour of sleep. Each patient will undergo three polysomnographic recordings (baseline, CPAP titration, after two months of treatment with oral appliance). Subjective (sleep disorders questionnaire, the Epworth Sleepiness Scale, and sleep diaries) and objective (polysomnography) parameters of sleep will be evaluated, besides the quality of life (SF-36), mood (POMS), and anthropometric measurements (neck circumference and craniofacial characteristic). Good response to treatment with the AIO will be considered as a 50% reduction in the baseline AHI index or AHI after treatment less than 5 events per hour of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 25 and 65 years old
* Epworth sleepiness Scale > 9
* Apnea-hypopnea index between 5 and 30

Exclusion Criteria:

* Presence of clinical disease (chronic obstructive pulmonary disease, asthma) and other sleep disorders.
* Presence of anatomical obstructive upper airway, tonsil grade III e IV, septal deviation and grade III that may affect the outcome of CPAP
* Loss of posterior dental support to undermine the retention of oral appliance
* Active of periodontal disease, compared Dental crow/dental root less than or equal to 1 (c/r ≤ 1) need primary dental care (cavities, root canal treatment or retreatment, dentures, i.e. outlying), open bite
* Protrusive displacement lass then five millimeters
* Limited mouth opening
* Alcoholism
* Use of sleep-inducing medications
* Habits or occupation that lead to sleep deprivation or alteration of the sleep-wake cycle
* Intolerance to CPAP
* Obesity grade II (moderate) or III (severe)

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Objective sleep parameters | two months after the baseline recording
  polysomnographic date of sleep stages percentages, sleep efficience, arousals, apnea-hypopnea index, oxyhemoglobin saturation

SECONDARY OUTCOMES:
Subjective sleep parameters | two months after the baseline recording
  Sleep disorders questionnaire, the Epworth Sleepiness Scale, and sleep diaries
Quality of life, mood, and anthropometric measurements | two months after the baseline recording
  SF-36, POMS, neck circumference and craniofacial characteristic

CONTACTS AND LOCATIONS:
Overall Officials: Lia Rita A Bittencourt, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Instituto do Sono/ Associação Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil